CLINICAL TRIAL: NCT02936804
Title: Key Technology in Precision Diagnosis and Therapy for Early Stage Lung Cancer: a Single Arm Clinical Trial
Brief Title: Precision Diagnosis and Therapy for Early Stage Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, : Vice-President, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chest002
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: early stage lung cancer; LDCT screening; lung resection; electromagnetic navigation bronchoscopy; peripheral biomarker
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening Arm (Experimental): Low Dose Computed Tomography (LDCT) was performed at baseline + 2 rounds of biennial repeated LDCT. Management of positive screening test will be carried out by a pre-specified protocol.
  Interventions: Device: Low Dose Computed Tomography

INTERVENTIONS:
Device: Low Dose Computed Tomography — LDCT was performed at baseline and 2 rounds of biennial repeated LDCT. The abnormal nodules were defined as noncalcified nodules (NCN) larger than 4 mm. The management of abnormal nodules including precision diagnosis by endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), electromagnetic navigation bronchoscope (ENB) and peripheral biomarkers, and precision therapy by intraoperative frozen section guided lung resection and ENB radiofrequency ablation.

SUMMARY:
The present study is a single arm clinical trial aiming to improve the key technology in the diagnosis and treatment of early stage lung cancer. 60,000 high-risk subjects (age 45-70) are planned to recruit and assign to the Low Dose Computed Tomography (LDCT) screening arm (Baseline + 2 rounds of biennial repeated LDCT screening). Management of positive screening test will be carried out by a pre-specified protocol.

ELIGIBILITY:
Inclusion Criteria:

• Eligible participants were those aged 45-70 years, and with either of the following risk factors:

1. history of cigarette smoking ≥ 20 pack-years, and, if former smokers, had quit within the previous 15 years;
2. malignant tumors history in immediate family members;
3. personal cancer history;
4. professional exposure to carcinogens;
5. long term exposure to second-hand smoke;
6. long term exposure to cooking oil fumes.

Exclusion Criteria:

1. Had a CT scan of chest within last 12 months
2. History of any cancer within 5 years

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60000 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Lung cancer incidence rate | 5 years
  Assess the number of lung cancer incidences after each round of screening. Compared the stage differences between screening arm and natural incidence.

SECONDARY OUTCOMES:
Lung cancer disease free survival | 5 years
  Compared the disease-free survival (DFS) among different treatment strategy of early stage lung cancer.
Lung cancer mortality | 5 years
  Assess lung cancer mortality within next 5 years after first round of screening

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided